CLINICAL TRIAL: NCT04749342
Title: Complete Decongestive Therapy Versus Compression Bandaging in Advanced Secondary Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mohamed Abdelrauf (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Abdelrauf, Complete Decongestive Therapy Versus Compression Bandaging in Advanced Secondary Lymphedema, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002271
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Edema Due to Obstruction of Lymph Vessels or Excision of Lymph Nodes

STUDY DESIGN:
Intervention Model Description: The purpose of this report is to compare short-term outcomes of complete decongestive therapy and compression bandaging on patients with advanced secondary upper and lower extremity lymphedema.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Decongestive Therapy (Experimental): Complete decongestive therapy (CDT) is also known as complex decongestive therapy. It involves a two-stage treatment protocol. The first stage consists of skin care, manual lymph drainage, exercises and compression with multi-layered bandages. The second stage aims to optimize and conserve the volume reduction obtained in stage one. This is achieved by using a low-stretch elastic garment in combination with skin care and exercises
  Interventions: Other: Physiotherapy Treatment
- Compression Bandaging (Experimental): External compression is the mainstay of management for all stages of lymphedema. The efficacy of compression therapy alone, or combined with MLD, has been supported by randomized clinical trials
  Interventions: Other: Physiotherapy Treatment

INTERVENTIONS:
Other: Physiotherapy Treatment — Physical Therapy sessions for treatment of advanced Lymphedema Cases

SUMMARY:
The purpose of this study is to:

Find out the efficacy of using complete decongestive physiotherapy on limb volume in advanced secondary upper and lower extremity lymphedema patients.

Find out the efficacy of compression bandaging on limb volume in advanced lymphedema patients.

This study was conducted to compare between the efficacy of complete decongestive therapy (CDT) and compression bandaging in advanced secondary lower extremity lymphedema.

DETAILED DESCRIPTION:
The study was conducted at the department of plastic surgery, Kasr Al-Ainy hospital. Sixty patients of both genders aged from 40 to 55 years old were participated in this study, and they were randomly assigned to two study groups.

Group I: Thirty patients received CDT (60 min of manual lymph drainage MLD, compression bandaging, exercises, and skin care).

Group II: Thirty patients received compression bandaging alone. The same bandaging scheme used for both groups. The therapy included 12 interventions performed 5 days a week, during the first two weeks in addition to another successive two sessions at the third week, i.e., for a total of twelve sessions.

Evaluation of limb volume using water volumetry and 4-cm truncated cone circumferential measurements were done before treatment application, after 6 sessions (post 1) and after 12 sessions (post 2).

ELIGIBILITY:
Inclusion Criteria:

Patients with lower limb lymphedema (stage II and III) secondary lymphedema aged from 40 to 55 years old, with BMI less than 35 and duration of illness ranged from 3-9 years were included in the study

Exclusion Criteria:

the patients were excluded if they have acute erysipelas, acute thrombophlebitis phlebothrombosis and decompensated heart failure.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Limb Volume | 1 Month
  girth Limb Measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Abdelrauf, Assistant Lecturer, Principal Investigator — Cairo University
Locations (1):
- cairo University, Cairo, Dokky, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
(all collected IPD, all IPD that underlie results in a publication)
Supporting Information: Study Protocol, SAP
Time Frame: Starting in December 2020 - March 2021